CLINICAL TRIAL: NCT00914589
Title: A Multi-Centre, Randomised, Double-Blind, Placebo Controlled Trial on Efficacy and Safety of FXIII Replenishment With Two Different Doses of Recombinant Factor XIII Following Cardiopulmonary Bypass Surgery
Brief Title: Multi-national Study Investigating the Effect and Safety of rFXIII on Transfusion Needs in Patients Undergoing Heart Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NN1810-3540; JapicCTI-101078 (Registry Identifier: JAPIC); 2008-006324-62 (EudraCT Number)
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Cardiac Surgery Requiring Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FXIII17.5IU/Kg (Experimental): Recombinant factor XIII at a single dose of 17.5 IU/kg lean body mass (LBM) was administered via slow i.v. push at a rate not exceeding two mL per minute.
  Interventions: Drug: catridecacog
- FXIII35IU/Kg (Experimental): Recombinant factor XIII at a single dose of 35 IU/kg lean body mass (LBM) was administered via slow i.v. push at a rate not exceeding two mL per minute.
  Interventions: Drug: catridecacog
- Placebo (Placebo Comparator): Recombinant factor XIII placebo was administered as a single dose via slow i.v. push at a rate not exceeding two mL per minute.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: catridecacog — Single dose via slow intravenous (i.v.) push at a rate not exceeding two mL per minute
  Arms: FXIII17.5IU/Kg
Drug: catridecacog — Single dose via slow intravenous (i.v.) push at a rate not exceeding two mL per minute
  Arms: FXIII35IU/Kg
Drug: placebo — Single dose via slow intravenous (i.v.) push at a rate not exceeding two mL per minute
  Arms: Placebo

SUMMARY:
This trial is conducted in Canada, Asia, Europe and USA. The aim of this clinical trial is to investigate the effect and safety of rFXIII on transfusion needs in patients undergoing heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* - Planned coronary artery bypass grafting (CABG) or CABG plus single heart valve replacement/repair or planned replacement/repair of a single heart valve

Exclusion Criteria:

* Known intolerance to protamine
* Known or suspected allergy to the used antifibrinolytic agent
* Refusal to receive blood or blood product
* Planned surgery including the aortic arch and/or descending aorta
* Planned surgery including any implantable ventricular assist device
* Adult congenital heart diseases
* Two or more previous cardiac surgery procedures
* Any known autoimmune diseases: Collagen vascular disease (Systemic lupus erythematosus, Rheumatoid arthritis, Sjögrens syndrome) - Endocrine: hyperthyroidism (Graves disease), adrenal insufficiency, Hashimoto's thyroiditis - Neurologic: Multiple sclerosis, myasthenia gravis - Skin: pemphigous vulgaris Hematologic: Pernicious anaemia, Autoimmune haemolytic anaemia - Vasculitis - Primary or secondary antiphospholipid syndrome
* Weight above 140 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (31):
- United States (7):
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Allentown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Providence, Rhode Island
  - Novo Nordisk Investigational Site, Houston, Texas
- Canada (5):
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal
  - Novo Nordisk Investigational Site, Ottawa
  - Novo Nordisk Investigational Site, Québec
  - Novo Nordisk Investigational Site, Toronto
- Novo Nordisk Investigational Site, København Ø, Denmark
- Germany (4):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Frankfurt am Main
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, München
- Israel (2):
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Ramat Gan
- Italy (3):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, San Donato Milanese (MI)
- Japan (3):
  - Novo Nordisk Investigational Site, Numakunai
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Tokyo
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Valencia
- Novo Nordisk Investigational Site, Lund, Sweden
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Southampton

REFERENCES:
- [Result] Song HK, von Heymann C, Jespersen CM, Karkouti K, Korte W, Levy JH, Ranucci M, Saugstrup T, Sellke FW. Safe application of a restrictive transfusion protocol in moderate-risk patients undergoing cardiac operations. Ann Thorac Surg. 2014 May;97(5):1630-5. doi: 10.1016/j.athoracsur.2013.12.025. Epub 2014 Mar 19. PMID 24655469
- [Derived] Karkouti K, von Heymann C, Jespersen CM, Korte W, Levy JH, Ranucci M, Sellke FW, Song HK. Efficacy and safety of recombinant factor XIII on reducing blood transfusions in cardiac surgery: a randomized, placebo-controlled, multicenter clinical trial. J Thorac Cardiovasc Surg. 2013 Oct;146(4):927-39. doi: 10.1016/j.jtcvs.2013.04.044. Epub 2013 Jun 29. PMID 23820174
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of a total of 32 initiated trial sites, 30 sites randomised and dosed at least one patient. The country distribution for these 30 sites was as follows (number of sites per country in parenthesis): Canada (5), Denmark (1), Germany (4), Great Britain (3), Israel (2), Italy (2), Japan (4), Spain (3) and the United States (6).
Pre-assignment Details: Seventy (70) of 479 subjects randomised in the trial were withdrawn before trial product administration.
Period: Overall Study
Arm/Group | Placebo | FXIII17.5IU/Kg | FXIII35IU/Kg
Started | 128 | 143 | 138
Completed | 103 | 127 | 126
Not Completed | 25 | 16 | 12
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Protocol Violation | 8 | 6 | 3
Not completed — unclassified | 16 | 9 | 7
Not completed — Death | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FXIII17.5IU/Kg | FXIII35IU/Kg | Total
Number analyzed (Participants) | 128 | 143 | 138 | 409
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (8.4) | 68.7 (9.0) | 69.0 (7.9) | 68.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 21 | 73
  Male | 100 | 119 | 117 | 336

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Avoiding Any Allogeneic Transfusions for Seven Days Post-operative or Until Discharge, Whichever Came First
Description: Proportion of patients avoiding blood products given via allogeneic transfusion. Blood products were defined as any of the following: RBC, platelets, FFP, fibrinogen concentrate and clotting factor(s) concentrate, including cryoprecipitate.
Time Frame: measured ongoing from dosing until day 7 or discharge, whichever came first
Population: Full analysis set consisted of all subjects who were randomised and exposed to randomised treatment.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Placebo | FXIII17.5IU/Kg | FXIII35IU/Kg
Number analyzed (Participants) | 128 | 143 | 138
percentage (%) of subjects
  Transfused | 35.2 | 35.7 | 34.1
  Not transfused | 64.8 | 64.3 | 65.9
Statistical Analysis 1: Comparison: Placebo vs FXIII17.5IU/Kg; Test type: Superiority or Other; p = 0.8648, Regression, Logistic — P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 1.0482, 95% CI [0.6095 to 1.8029]
Statistical Analysis 2: Comparison: Placebo vs FXIII35IU/Kg; Test type: Superiority or Other; p = 0.9634, Regression, Logistic — P values less than 0.05 are considered statistically significant in this study; Odds Ratio (OR) = 0.9871, 95% CI [0.5673 to 1.7176]

2. Secondary Outcome: Percentage of Subjects With Thromboembolic Events
Description: Percentage of subjects with thromboembolic events (AMI, cerebrovascular thromboembolic event, peripheral artery occlusion, DVT, pulmonary embolism) until end of trial
Time Frame: measured from screening until 5-7 weeks post Trial Drug Administration
Population: The safety analysis set included all subjects who were exposed to at least one dose of trial product.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | FXIII17.5IU/Kg | FXIII35IU/Kg
Number analyzed (Participants) | 128 | 143 | 138
percentage of subjects
  All events | 9.38 | 8.39 | 6.52
  Peri-operative Acute Myocardial infarcti | 6.25 | 6.99 | 5.07
  Cerebrovascular Thromboembolic Event | 2.34 | 1.40 | 0.00
  Deep vein thrombosis | 0.78 | 0.00 | 0.72
  Peripheral Artery Occlusion | 0.00 | 0.00 | 0.72

3. Secondary Outcome: Percentage of Subjects With rFXIII Antibody Reaction
Description: Immunogenicity as number of subjects who manifested FXIII antibody reaction until end of trial. The percentage may be derived from the number of subjects treated with rFXIII with available antibody measurement at visit 8.
Time Frame: measured from screening until 5-7 weeks post Trial Drug Administration
Population: Safety analysis set includes all subj. exposed to at least one dose of trial product. 1 subj with a low titre antibody at baseline was also reported with low titre FXIII antibody at visit 8. 27, 19 and 17 subjects in placebo, FXIII 17.5 and 35 IU/KG, respectively, did not have antibody measurement.
Measure: Number; unit: participants
Arm/Group | Placebo | FXIII17.5IU/Kg | FXIII35IU/Kg
Number analyzed (Participants) | 101 | 124 | 121
participants | 0 | 1 | 0

4. Secondary Outcome: Percentage of Subjects With Critical Adverse Events
Description: Percentage of subjects with critical adverse events (thromboembolic events (AMI, cerebrovascular thromboembolic event, peripheral artery occlusion, DVT, pulmonary embolism), renal dysfunction, re-operation and death) until end of trial
Time Frame: measured from screening until 5-7 weeks post Trial Drug Administration
Population: The safety analysis set included all subjects who were exposed to at least one dose of trial product.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Placebo | FXIII17.5IU/Kg | FXIII35IU/Kg
Number analyzed (Participants) | 128 | 143 | 138
percentage (%) of subjects
  All events | 14.84 | 16.78 | 11.59
  Peri-operative Acute Myocardial Infarcti | 6.25 | 6.99 | 5.07
  Renal dysfunction | 7.03 | 6.99 | 3.62
  Re-operation | 1.56 | 5.59 | 2.90
  Cerebrovascular Thromboembolic Event | 2.34 | 1.40 | 0.00
  Death | 0.00 | 0.70 | 0.72
  Deep vein thrombosis | 0.78 | 0.00 | 0.72
  Peripheral artery Occlusion | 0.00 | 0.00 | 0.72

5. Secondary Outcome: Percentage of Subjects With Serious Adverse Events
Description: Percentage of subjects with serious adverse events until end of trial.
Time Frame: measured from screening until 5-7 weeks post Trial Drug Administration
Population: The safety analysis set included all subjects who were exposed to at least one dose of trial product.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Placebo | FXIII17.5IU/Kg | FXIII35IU/Kg
Number analyzed (Participants) | 128 | 143 | 138
percentage (%) of subjects
  Blood and lymphatic system disorders | 0.00 | 0.70 | 0.00
  Cardiac disorders | 8.59 | 12.59 | 7.25
  Eye disorders | 0.00 | 0.70 | 0.00
  Gastrointestinal disorders | 1.56 | 0.70 | 0.00
  General disorders and administration sit | 1.56 | 0.00 | 2.17
  Infections and infestations | 5.47 | 5.59 | 3.62
  Injury, poisoning and procedural compli | 2.34 | 4.90 | 2.90
  Investigations | 0.00 | 0.00 | 0.72
  Musculoskeletal and connective tissue d | 0.00 | 0.70 | 0.00
  Neoplasms benign, malignant and unspecif | 0.78 | 0.00 | 0.00
  Nervous system disorders | 3.91 | 2.80 | 2.17
  Psychiatric disorders | 0.00 | 0.70 | 0.72
  Renal and urinary disorders | 1.56 | 2.10 | 2.17
  Respiratory, thoracic and mediastinal d | 7.03 | 6.29 | 7.25
  Skin and subcutaneous tissue disorders | 0.78 | 0.00 | 0.00
  Vascular disorders | 1.56 | 1.40 | 1.45

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of rFXIII dosing until day 7 or discharge (whichever came first), while serious adverse events were reported from the time of rFXIII dosing until the follow-up visit at 5-7 weeks after trial drug administration.
Description: Safety analysis set were all subjects who have been exposed to at least one dose of trial drug
Arm/Group | Placebo | FXIII17.5IU/Kg | FXIII35IU/Kg
Serious Adverse Events (participants affected / at risk) | 35/128 | 43/143 | 32/138
Other Adverse Events (participants affected / at risk) | 120/128 | 129/143 | 128/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=128) | FXIII17.5IU/Kg (N=143) | FXIII35IU/Kg (N=138)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 3 (3) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dressler (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal ischaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Graft dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Postoperative thoracic procedure comp (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Reversible ischaemic neurological def. (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 2 (2)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=128) | FXIII17.5IU/Kg (N=143) | FXIII35IU/Kg (N=138)
Anaemia (Blood and lymphatic system disorders) | 25 (25) | 24 (25) | 19 (19)
Leukocytosis (Blood and lymphatic system disorders) | 9 (9) | 6 (6) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (11) | 5 (5) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 50 (56) | 45 (48) | 44 (49)
Low cardiac output syndrome (Cardiac disorders) | 9 (9) | 3 (3) | 10 (10)
Ventricular extrasystoles (Cardiac disorders) | 6 (6) | 4 (4) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6) | 6 (6) | 9 (9)
Nausea (Gastrointestinal disorders) | 34 (34) | 38 (38) | 46 (46)
Vomiting (Gastrointestinal disorders) | 10 (13) | 15 (15) | 21 (21)
Chills (General disorders) | 12 (12) | 5 (5) | 8 (8)
Oedema peripheral (General disorders) | 18 (19) | 23 (27) | 25 (28)
Pyrexia (General disorders) | 17 (17) | 15 (15) | 14 (15)
Anaemia postoperative (Injury, poisoning and procedural complications) | 8 (8) | 7 (7) | 8 (9)
Procedural pain (Injury, poisoning and procedural complications) | 34 (35) | 45 (47) | 45 (47)
Wound secretion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 10 (10)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 8 (8) | 3 (3)
Urine output decreased (Investigations) | 9 (9) | 9 (9) | 9 (9)
Fluid overload (Metabolism and nutrition disorders) | 11 (11) | 10 (10) | 15 (15)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (16) | 19 (19) | 21 (21)
Hypovolaemia (Metabolism and nutrition disorders) | 12 (12) | 12 (12) | 7 (7)
Dizziness (Nervous system disorders) | 4 (4) | 8 (9) | 9 (9)
Agitation (Psychiatric disorders) | 8 (9) | 5 (5) | 4 (4)
Delirium (Psychiatric disorders) | 10 (10) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 9 (10) | 10 (11) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 15 (16) | 13 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 9 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 48 (50) | 42 (45) | 52 (54)
Hypertension (Vascular disorders) | 5 (5) | 5 (5) | 13 (13)
Hypotension (Vascular disorders) | 28 (29) | 17 (17) | 21 (22)
Haemorrhage (Vascular disorders) | 4 (4) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.